CLINICAL TRIAL: NCT05317949
Title: Effect of Integrated Neuromuscular Training on Explosive Strength, Speed and Endurance of Medium Fast Bowler in Cricket
Brief Title: Effect of Integrated Neuromuscular Training on Medium Fast Bowler in Cricket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01254 Nadeem Afsar
Record Dates: First submitted 2022-04-02; First posted 2022-04-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sports Physical Therapy
Keywords: Sports Rehabilitation; Integrated Neuromuscular Training; Speed; Endurance; Explosive strength; Fast bowler; Cricket

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated neuromuscular training program group (Experimental): Integrated neuromuscular training program group will perform exercise in three major domains
  Interventions: Other: Integrated neuromuscular training program group
- General fitness exercises program group (Active Comparator): General fitness exercises program group will perform general fitness exercises
  Interventions: Other: General fitness exercises program group

INTERVENTIONS:
Other: Integrated neuromuscular training program group — Integrated neuromuscular training program group will do plyometric training, speed and sensitivity training, resistance training for 3 days in a week and total for eight weeks.
  Arms: Integrated neuromuscular training program group
Other: General fitness exercises program group — General fitness exercises program group will do general fitness exercise for 3 days in a week and total for eight weeks.
  Arms: General fitness exercises program group

SUMMARY:
Effect of Integrated Neuromuscular Training on Explosive Strength, Speed and Endurance of Medium Fast Bowler in Cricket

DETAILED DESCRIPTION:
Integrated neuromuscular training (INT) is a combination of functional movement training and speciﬁc strength, balance, speed, sensitivity, and isometric training, which aims to evaluate and prevent sports injury and improve sports performance. Neuromuscular control defects are mainly manifested as decreases in muscle strength, explosive power, or abnormal activation patterns. INT is deﬁned as a conceptual training program that incorporates general (e.g., fundamental movements) and speciﬁc strength and conditioning tasks (e.g., resistance, balance, agility, plyometric) to improve injury resilience and to enhance sporting and motor skill performance. The majority of studies in youth examining neuromuscular training strategies to improve performance and injury prevention include multiple components (for example, balance, strength, plyometric, agility, speed, coordination. INT sessions are characterized by short bursts of physical activity interspersed with brief rest periods.

the purpose of this study is to find the effect of integrated neuromuscular training on explosive strength, speed and endurance of medium fast bowler in cricket

ELIGIBILITY:
Inclusion Criteria:

* Medium fast bowlers
* Players playing cricket for > 1 year
* Players engaging in cricket ≥ 3 days in a week

Exclusion Criteria:

* History of any injury in past 6 months.
* Those players having musculoskeletal, neurological, cardiorespiratory problems
* Those players who have any medical condition

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Soft Ball Throw Test | Eight weeks
  the test involves throwing a soft for maximum distance this test measure explosive power, particularly of the upper body and evaluate throwing distance
50 Yard Dash | Eight weeks
  The aim of this test is to determine acceleration and speed procedure : The test involves running a single maximum sprint over 50 meters, with the time recorded.
1 Mile Run Test | Eight weeks
  The purpose of this test is to complete one mile in the fastest possible time. After the purpose of the test and instructions are given, the participants begin running on the count "Ready? Go!"

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, Ph.D*, Principal Investigator — Riphah International University
Locations (1):
- Sports Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No